CLINICAL TRIAL: NCT03931174
Title: Implementing Contingency Management in Opioid Treatment Centers Across New England: A Type 3 Hybrid Trial
Brief Title: Project MIMIC (Maximizing Implementation of Motivational Incentives in Clinics)
Acronym: MIMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: RTI International (Other); University of Washington (Other); UConn Health (Other); National Institute on Drug Abuse (NIDA) (NIH); Northwestern University (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: #1811002260; R01DA046941 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder
Keywords: implementation; opioid use
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addiction Technology Transfer Center (ATTC) Training (Active Comparator): Half of the opioid treatment centers will receive the ATTC training strategy.
  Interventions: Behavioral: Addiction Technology Transfer Center (ATTC) Training Strategy
- Enhanced ATTC (E-ATTC) Training Strategy (Experimental): Half of the opioid treatment centers will receive the E-ATTC training strategy.
  Interventions: Behavioral: Enhanced Addiction Technology Transfer Center (E-ATTC) Training Strategy

INTERVENTIONS:
Behavioral: Addiction Technology Transfer Center (ATTC) Training Strategy — Participating organizations will receive training consisting of 3 components: 1) didactic workshop - full-day workshop led by a contingency management (CM) expert for both CM staff and leaders, 2) performance feedback - submission of CM session recordings for review and performance feedback at least monthly for 9 months for CM staff, and 3) staff coaching - monthly provider coaching calls led by a CM expert for 9 months for both CM staff and leaders.
  Other Names: ATTC
  Arms: Addiction Technology Transfer Center (ATTC) Training
Behavioral: Enhanced Addiction Technology Transfer Center (E-ATTC) Training Strategy — Participating organizations will receive all of the elements of the ATTC control condition. In addition, organizations will receive two additional elements: 1) Implementation Sustainment Facilitation - monthly coaching calls for CM leaders and staff focused on sustainment, 2) Pay for Performance - participating CM staff will have the opportunity to earn monthly monetary bonuses for achieving pre-defined implementation goals for 9 months.
  Other Names: E-ATTC
  Arms: Enhanced ATTC (E-ATTC) Training Strategy

SUMMARY:
There is an urgent need for effective treatments for patients with opioid use disorder (OUD). This study will train opioid treatment programs in an evidence-based behavioral treatment called contingency management (CM). Contingency management (i.e., motivational incentives for achieving pre-defined treatment goals) is one of the only behavioral interventions shown to improve patient treatment outcomes when combined with FDA-approved pharmacotherapy. Unfortunately, however, uptake of CM in opioid treatment programs remains low. In response to the urgent need for evidence-based behavioral OUD treatments, the investigators propose a large-scale type 3 hybrid trial comparing two comprehensive strategies to promote CM implementation as an adjunct to pharmacotherapy within opioid treatment programs. The control condition is the staff training strategy used by the New England Addiction Technology Transfer Center, which consists of didactic workshop, performance feedback, and staff coaching. The experimental condition is the ATTC strategy enhanced by external leadership coaching (using a model called Implementation Sustainment Facilitation; ISF) and provider incentives (using a model called Pay for Performance; P4P).

A cluster randomized design trial will be conducted with 30 opioid treatment programs across New England. Centers will be randomized to one of the two implementation conditions (ATTC vs. enhanced-ATTC) over the 5 year project. At each opioid treatment program, data will be collected at multiple intervals from CM treatment providers, organizational leaders, and newly admitted patients. Additionally, patient charts will be randomly selected for review to examine sustainment. Data collection will include electronic medical record review, ratings of audio recordings by staff blind to condition, well-validated measures, and provider weekly report of patient encounter data. Specific Aims of the study are to experimentally compare the effect of the two conditions on implementation outcomes (Primary Aim) and on patient outcomes (Secondary Aim). An Exploratory Aim is to test whether two organization-level variables (i.e., implementation climate, leadership engagement) partially mediate the relationship between implementation condition and the key study outcomes.

DETAILED DESCRIPTION:
Overdoses and deaths due to opioid use disorders (OUDs) have been declared a public health emergency in the United States, bringing to light an urgent need for highly effective OUD treatments. There are currently five FDA-approved medication formulations, which relative to placebo have demonstrated effectiveness in helping patients attain abstinence from opioids. Nonetheless, patients' opioid abstinence rates are sub-optimal: even when treated with the newest extended-release formulations only about 40% of patients maintain abstinence during the first 6-months of treatment. Contingency management (CM; i.e., motivational incentives for achieving pre-defined treatment goals) is one of the only behavioral interventions shown to improve patient abstinence from opioids when combined with FDA-approved pharmacotherapy. Unfortunately, however, uptake of CM in opioid treatment programs remains low.

The primary purpose of this study is to experimentally evaluate two different comprehensive training models to train opioid treatment programs in CM. A Type 3 Hybrid Trial will be conducted collecting data on both implementation and patient outcomes. Using a cluster randomized design, 30 opioid treatment programs across New England will be randomized to one of two comprehensive training conditions over a 5 year period. The control condition is the staff training strategy used by the Substance Abuse and Mental Health Services Administration (SAMHSA)-funded network of Addiction Technology Transfer Centers (ATTC; i.e., didactic workshop + performance feedback + staff coaching). The experimental condition is the ATTC strategy enhanced by external leadership coaching (using a model called Implementation Sustainment Facilitation [ISF], i.e., leadership coaching focused on sustainment planning) and provider incentives (using a model called Pay for Performance [P4P]; i.e., monetary bonuses for achieving pre-defined implementation goals), hereafter referred to as E-ATTC. Elements of the E-ATTC condition were informed by our team's prior NIH-funded work evaluating organization-level implementation strategies. At each OUD treatment center, data will be collected at multiple intervals from up to 2-5 CM treatment providers (n=60-150 providers), 1-2 organizational leaders (n=30-60 leaders), and 25 newly admitted patients (n=750 patients). Additionally, 25 patient charts per center (n=750 charts) will be randomly selected for review to examine sustainment. Data collection will include electronic medical record review, ratings of audio recordings by staff blind to condition, well-validated measures, and biological verification of abstinence.

The Primary Aim of the study is to experimentally compare the effect of the two training strategies on implementation outcomes. Focal implementation outcomes include: CM Exposure (provider-level measure of the proportion of providers delivering the target number of CM sessions to at least one patient during 9-month Implementation phase), CM Competence (provider-level measure of CM quality during month Implementation phase), and CM Sustainment (organization-level measure of the proportion of programs continuing to deliver CM sessions during 6-month Sustainment phase).

The Secondary Aim of the study is to experimentally compare the effect of the two training strategies on patient outcomes. Focal patient outcomes include abstinence from opioids and opioid-related problems.

An Exploratory Aim is to test whether two provider-level variables (i.e., implementation climate, leadership engagement) partially mediate the relationship between implementation condition and the key study outcomes.

Pursuit of these aims is significant given the potential to improve the treatment of OUDs in community settings, which is one of the greatest public health challenges currently facing our nation. Major strengths of the approach include the study's experimental design (cluster randomized trial), novel implementation strategy based on mixed-methods pilot data by the investigative team, large sample of organizations (N = 30), partnership with a SAMHSA-funded national training center, and rigorously measured implementation and patient outcomes.

ELIGIBILITY:
Inclusion criteria for community-based opioid treatment programs (n = 30):

* prescribes FDA-approved medication to treat adult patients with OUDs
* enrolls 5+ new patients per month
* has at least 2 staff who provide psychosocial support to OUD patients

Exclusion criteria:

• None

Inclusion criteria for CM Providers (n = 60-150, range of 2-5 per center):

* has been involved in providing psychosocial support to OUD patients on pharmacotherapy
* has an active caseload
* is willing to commit to 14 months of CM training and support

Exclusion criteria:

• None

Inclusion Criteria for CM Leaders (n = 30-60, range of 1-2 per center):

* is responsible for supervising frontline CM Staff
* is willing to commit to 14 months of external leadership coaching

Exclusion criteria:

• None

Inclusion criteria for patients (n = 750):

* adult patients
* newly admitted to the opioid treatment center within the past 30 days
* prescribed any FDA-approved OUD medication

Exclusion criteria:

• issues that could interfere with the ability to complete a brief intake interview including acute intoxication, acute psychosis, acute mania, or cognitive impairment (prohibiting comprehension of the consent process), as reported by opioid treatment program staff or observed by research staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Becker, Ph.D., Principal Investigator — Brown University and Northwestern University; Bryan R Garner, Ph.D., Principal Investigator — Ohio State University
Locations (29):
- United States (29):
  - Kinsella Treatment Center, Bridgeport, Connecticut
  - Liberation Programs Bridgeport, Bridgeport, Connecticut
  - Community Renewal Team, Hartford, Connecticut
  - Liberation Programs Stamford, Stamford, Connecticut
  - North Charles Institute for the Addictions, Cambridge, Massachusetts
  - Habit Opco East Wareham Comprehensive Treatment Center, East Wareham, Massachusetts
  - Habit Opco Fall River Comprehensive Treatment Center, Fall River, Massachusetts
  - Spectrum Health Systems Framingham, Framingham, Massachusetts
  - Spectrum Health Systems Haverhill, Haverhill, Massachusetts
  - Spectrum Health Systems Leominster, Leominster, Massachusetts
  - Spectrum Health Systems Milford, Milford, Massachusetts
  - Spectrum Health Systems Millbury, Millbury, Massachusetts
  - Gifford Street Comprehensive Treatment Center, New Bedford, Massachusetts
  - Spectrum Health Systems North Adams, North Adams, Massachusetts
  - Spectrum Health Systems Pittsfield, Pittsfield, Massachusetts
  - Spectrum Health Systems Southbridge, Southbridge, Massachusetts
  - Habit Opco Taunton Comprehensive Treatment Center, Taunton, Massachusetts
  - Spectrum Health Systems Waltham, Waltham, Massachusetts
  - Spectrum Health Systems Weymouth, Weymouth, Massachusetts
  - Spectrum Health Systems Worcester, Worcester, Massachusetts
  - Habit Opco West Lebanon Comprehensive Treatment Center, West Lebanon, New Hampshire
  - CODAC Behavioral Healthcare - Eleanor Slater, Cranston, Rhode Island
  - Lifespan Recovery Center, Providence, Rhode Island
  - Discovery House Comprehensive Treatment Center, Providence, Rhode Island
  - VICTA, Providence, Rhode Island
  - CODAC Providence, Providence, Rhode Island
  - Woonsocket Comprehensive Treatment Center, Woonsocket, Rhode Island
  - BAART Programs Berlin, Berlin Corners, Vermont
  - West Ridge Center, Rutland, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan for the primary outcomes has been published in Addiction Science and Clinical Practice. Additional data (analytic code, participant-level data) can be requested from the Multiple Principal Investigators. Analysis files will be constructed from the stored electronic data and will be stripped of identifying information. Specifically, participants will be identified with a numeric identifier that is not related to any element of their personal identifying information. No names, addresses, telephone numbers, fax numbers, email addresses, social security numbers, medical records, etc. will be retained.
Supporting Information: Study Protocol, SAP
Time Frame: Protocol was published in 2021. Analytic code and participant-level data were made ready for distribution by July 30, 2024.
Access Criteria: Data will only be shared with external investigators when a data use agreement (DUA) is executed between Brown University and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project, and schedule for data destruction.

REFERENCES:
- [Derived] Becker SJ, Janssen T, Murphy CM, Scott K, DiClemente-Bosco K, Souza T, Garner BR. Project MIMIC (Maximizing Implementation of Motivational Incentives in Clinics): preparation phase outcomes of a hybrid type 3 trial. Implement Sci Commun. 2025 Dec 15. doi: 10.1186/s43058-025-00841-7. Online ahead of print. PMID 41398966
- [Derived] Becker SJ, Janssen T, Souza T, Hartzler B, Rash CJ, DiClemente-Bosco K, Garner BR. Project MIMIC (Maximizing Implementation of Motivational Incentives in Clinics): results of a 28-site cluster-randomized type 3 hybrid trial. Implement Sci. 2025 Dec 9;21(1):9. doi: 10.1186/s13012-025-01473-0. PMID 41361474
- [Derived] Frohe T, Janssen T, Garner BR, Becker SJ. Examining changes in pain interference via pandemic-induced isolation among patients receiving medication for opioid use disorder: a secondary data analysis. BMC Public Health. 2024 Sep 27;24(1):2581. doi: 10.1186/s12889-024-20077-9. PMID 39334184
- [Derived] Janssen T, Garner BR, Yermash J, Yap KR, Becker SJ. Early COVID-Related pandemic impacts and subsequent opioid outcomes among persons receiving medication for opioid use disorder: a secondary data analysis of a Type-3 hybrid trial. Addict Sci Clin Pract. 2023 Sep 13;18(1):54. doi: 10.1186/s13722-023-00409-7. PMID 37705105
- [Derived] Becker SJ, Murphy CM, Hartzler B, Rash CJ, Janssen T, Roosa M, Madden LM, Garner BR. Project MIMIC (Maximizing Implementation of Motivational Incentives in Clinics): A cluster-randomized type 3 hybrid effectiveness-implementation trial. Addict Sci Clin Pract. 2021 Oct 12;16(1):61. doi: 10.1186/s13722-021-00268-0. PMID 34635178

RESULTS

PARTICIPANT FLOW:
Period: Providers
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Started (Referred to as Baseline in our analysis) | 95 | 91
Midpoint of Active Implementation (4.5 Months Post Baseline) | 62 (Completed N=62 (95%) ATTC out of 65 Active) | 63 (Completed N=63 (100%) E-ATTC out of 63 Active)
Endpoint of Active Implementation (9 Months Post Baseline) | 54 (Completed N=54 (93%) ATTC out of 58 Active) | 58 (Completed N=58 (94%) E-ATTC out of 62 Active)
Completed | 54 | 58
Not Completed | 41 | 33
Not completed — Staff left organization | 26 | 25
Not completed — Staff on leave/no longer engaged in implementation initiative | 11 | 4
Not completed — Lost to Follow-up | 4 | 4
Period: Patients
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Started (Referred to as Baseline in our analysis) | 286 | 308
3-month Follow-up | 225 (Completed N=225 (79.2%) ATTC out of 284 Active) | 240 (Completed N=240 (78.4%) E-ATTC out of 306 Active)
6-month Follow-up | 224 (Completed N=224 (78.9%) ATTC out of 284 Active) | 217 (Completed N=217 (70.9%) E-ATTC out of 306 Active)
Completed | 224 | 217
Not Completed | 62 | 91
Not completed — Post-consent screening failure | 1 | 1
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 60 | 89

BASELINE CHARACTERISTICS:
Population: These numbers include both providers (95= ATTC, 91= E-ATTC) and patients (286= ATTC, 308= E-ATTC)
Groups:
- Total: Total of all reporting groups
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy | Total
Number analyzed (Participants) | 381 | 399 | 780
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: Age was assessed by provider (95= ATTC, 91= E-ATTC) and patient (286= ATTC, 308= E-ATTC) groups.
  Years
    Providers: number analyzed (Participants) | 95 | 91 | 186
    Providers | 40.92 (12.56) | 38.68 (12.21) | 39.83 (12.40)
    Patients: number analyzed (Participants) | 286 | 308 | 594
    Patients | 38.15 (10.11) | 37.48 (10.28) | 37.83 (10.19)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/Gender was assessed by provider (95= ATTC, 91= E-ATTC) and patient (286= ATTC, 308= E-ATTC) groups.
  Participants
    Providers: number analyzed (Participants) | 95 | 91 | 186
    Providers: Female | 77 | 75 | 152
    Providers: Male | 18 | 16 | 34
    Patients: number analyzed (Participants) | 286 | 308 | 594
    Patients: Female | 129 | 137 | 266
    Patients: Male | 157 | 171 | 328
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity was assessed by provider (95= ATTC, 91= E-ATTC) and patient (286= ATTC, 308= E-ATTC) groups.
  Participants
    Providers: number analyzed (Participants) | 95 | 91 | 186
    Providers: American Indian or Alaska Native | 1 | 0 | 1
    Providers: Asian | 1 | 0 | 1
    Providers: Native Hawaiian or Pacific Islander | 0 | 0 | 0
    Providers: Black or African American | 6 | 7 | 13
    Providers: White | 74 | 73 | 147
    Providers: More than one race | 9 | 8 | 17
    Providers: Unknown or Not Reported | 4 | 3 | 7
    Patients: number analyzed (Participants) | 286 | 308 | 594
    Patients: American Indian or Alaska Native | 3 | 5 | 8
    Patients: Asian | 0 | 4 | 4
    Patients: Native Hawaiian or Pacific Islander | 2 | 1 | 3
    Patients: Black or African American | 20 | 22 | 42
    Patients: White | 212 | 233 | 445
    Patients: More than one race | 20 | 15 | 35
    Patients: Unknown or Not Reported | 29 | 28 | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Providers | 95 | 91 | 186
  United States: Patients | 286 | 308 | 594
CM Exposure [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: CM Exposure (Implementation Outcome)
Description: Provider-level measure of whether the provider delivered the target number of CM sessions (at least 10 sessions) to at least one patient based on based on electronic medical record review and data entered into a study-specific CM tracker tool for up to 25 charts per site (25 charts*30 sites = 750 charts). Providers will report on patient encounters in the electronic medical record and the study-specific CM tracker tool, and for each encounter will report if CM was provided. Using patient level data, providers will be classified as 1 (delivered 10 or more sessions to at least 1 patient) or 0 (did not deliver 10 or more CM sessions to any patients).
  *This measure was initially defined as a patient-level outcome. We altered the level at which CM Exposure was assessed because our initial approach excluded providers who were trained but never delivered CM. To follow intent-to-treat principles, we aggregate CM Exposure data at the provider-level in a manner that uses all available data.
Time Frame: From baseline to 9 months post-baseline
Population: Table reports proportions with listwise deletion. The pre-specified plan uses mixed models with full maximum likelihood estimation (intent-to-treat) and data from all 95 ATTC providers and 91 E-ATTC.
Measure: Count of Participants; unit: Participants
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Number analyzed (Participants) | 95 | 91
Participants | 18 | 31
Statistical Analysis 1: Comparison: Addiction Technology Transfer Center (ATTC) Training vs Enhanced ATTC (E-ATTC) Training Strategy; These analyses are unadjusted. The primary outcomes paper will report both unadjusted and adjusted analyses; Test type: Superiority — Unit of analysis is the provider level. All 186 providers (95 ATTC, 91 E-ATTC) who enrolled in the study are included in the analysis; p = 0.097, Mixed Models Analysis — CM Exposure is reported as the estimated proportion of providers delivering 10 or more CM sessions to at least one patient in a mixed model accounting for nesting; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.85 to 6.81], Standard Error of Mean 0.53

2. Primary Outcome: Contingency Management Competence Scale for Reinforcing Attendance (Implementation Outcome)
Description: Provider scores on the Contingency Management Competence Scale for Reinforcing Attendance (CMCS; Petry & Ledgerwood, 2010). Coders blind to treatment condition rate audio recorded CM sessions using the CMCS, which measures provider skill in CM delivery. CMCS contains 6 CM-specific skill items and 3 general skill items that are scored on a scale from 0 to 7. For each item, a score of 0 indicates an audio recording was not submitted, a score of 1 indicates the lowest possible skill and a score of 7 indicates the highest possible skill. Possible scale scores range from a minimum of 0 to 63. An average score will be calculated for each provider, with a minimum of 0 and maximum of 7. Providers will submit one audio recording per month for the duration of the 9-month Implementation phase. Each provider's highest CMCS score will be used in analysis. Higher scores indicate higher skill, which is a better outcome.
Time Frame: From baseline to 9 months post-baseline
Population: Table reports means and standard deviations. The pre-specified plan uses mixed models with full maximum likelihood estimation (intent-to-treat) and data from all 95 ATTC providers and 91 E-ATTC providers.
Measure: Mean (Standard Deviation); unit: Units on the CM Competence Scale
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Number analyzed (Participants) | 95 | 91
Units on the CM Competence Scale | 0.53 (1.66) | 1.25 (2.14)
Statistical Analysis 1: Comparison: Addiction Technology Transfer Center (ATTC) Training vs Enhanced ATTC (E-ATTC) Training Strategy; These analyses are unadjusted. The primary outcomes paper will report both unadjusted and adjusted analyses; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.02, t-test, 2 sided; T-test adjusted for inequality of variances; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [0.11 to 1.32], Standard Error of Mean 0.31

3. Primary Outcome: CM Sustainment (Implementation Outcome)
Description: Proportion of programs delivering any CM after removal of active support. This is calculated based on review of all patient charts over a 6-month interval. Providers report on patient encounters in the medical record, and for each encounter report if CM was provided. Programs are classified as 1 (reported delivering CM to at least 1 patient) or 0 (did not deliver CM to any patients). The proportion of programs delivering CM is then calculated; a higher proportion is a better outcome.
  *The level at which CM Sustainment was assessed was altered from provider-level to program-level because of the frequency of programs failing to report applying CM among any patients, across any of its providers. In addition, there was such high staff turnover we could not assess at the provider-level using original provider IDs. To be able to use all available data from all programs' medical records, we report on the proportion of any programs delivering CM after removal of active support.
Time Frame: 6-month time interval following Implementation time period
Population: Sustainment was measured at the organizational level (N=14 ATTC, N=14 E-ATTC) as a dichotomous variable indicating whether or not they continued delivering the intervention. The number of participants seen in each condition is unknown and therefore overall number of participants is entered as NA (not applicable).
Measure: Count of Units; unit: Organization Sites
Units Other Than Participants: Organization Sites
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Number analyzed (Participants) | NA | NA
Number analyzed (Organization Sites) | 14 | 14
Organization Sites | 6 | 6
Statistical Analysis 1: Comparison: Addiction Technology Transfer Center (ATTC) Training vs Enhanced ATTC (E-ATTC) Training Strategy; These analyses are unadjusted; Test type: Superiority — Unit of analysis is the organization-level. Total number of organizations included in the analysis is 28 (14 ATTC, 14 E-ATTC); p = 0.430, Chi-squared; Pearson Chi-Square; Chi-square test statistic value = 0.662

4. Secondary Outcome: Opioid Abstinence: Past Month (Patient Outcome)
Description: Days of abstinence as reported using calendar-based recall based on the Timeline Followback Interview method (Sobell & Sobell, 1992). Days of opioid abstinence will be calculated from 0 to 30 for each patient, with higher numbers indicating more days of abstinence (which is a better outcome). This will be calculated for all patients who complete follow-up.
Time Frame: Assessed at 3 and 6-months from patient baseline assessment
Population: Table reports means and standard deviations with listwise deletion. The pre-specified plan uses mixed models with full maximum likelihood estimation (intent-to-treat) and data from all patients who reported any follow-up data (N = 592).
Measure: Mean (Standard Deviation); unit: Days of opioid abstinence
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Number analyzed (Participants) | 286 | 308
Days of opioid abstinence
  3-months post baseline: number analyzed (Participants) | 226 | 236
  3-months post baseline | 8.89 (13.12) | 9.39 (14.00)
  6-months post baseline: number analyzed (Participants) | 223 | 217
  6-months post baseline | 10.15 (16.33) | 8.33 (14.70)
Statistical Analysis 1: Comparison: Addiction Technology Transfer Center (ATTC) Training vs Enhanced ATTC (E-ATTC) Training Strategy; These analyses are unadjusted. The primary outcomes paper will report both unadjusted and adjusted analyses; Test type: Superiority — Analyses are at the patient-level. All patients who enrolled in the study are included in the analysis; p = .034, Mixed Models Analysis; Mean Difference (Final Values) = -0.695, 95% CI 2-sided [-1.30 to -0.08], Standard Error of Mean 0.313

5. Secondary Outcome: Global Appraisal of Individual Needs Opioid-Related Problem Scale: Past Month (Patient Outcome)
Description: Count of problems as reported using an adapted version of the Global Appraisal of Needs Substance Problems Scale (Dennis et al., 2002), which has been adapted to focus specifically on problems related to opioids. The scale contains 16 items that correspond to problems related to opioid use. Patients are asked the last time they had each problem with responses including past month, past year, lifetime, or never. A count of problems experienced over the past month will be calculated for each patient. The minimum possible score is 0 and the maximum possible score is 16. Higher scores indicate higher problems, which is a worse outcome. This will be calculated for all patients who complete follow-up.
Time Frame: Assessed at 3 and 6-months from patient baseline assessment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Number analyzed (Participants) | 286 | 308
Units on a scale
  3-months post baseline: number analyzed (Participants) | 225 | 238
  3-months post baseline | 2.43 (3.51) | 2.55 (3.67)
  6-months post baseline: number analyzed (Participants) | 223 | 216
  6-months post baseline | 2.24 (3.47) | 2.17 (3.69)
Statistical Analysis 1: Comparison: Addiction Technology Transfer Center (ATTC) Training vs Enhanced ATTC (E-ATTC) Training Strategy; These analyses are unadjusted. The primary outcomes paper will report both unadjusted and adjusted analyses; Test type: Superiority — Analyses are at the patient-level. All patients who enrolled in the study are included in the analysis; p = 0.27, Mixed Models Analysis; Mean Difference (Final Values) = -0.202, 95% CI 2-sided [-0.82 to 0.41], Standard Error of Mean 0.314

6. Other Pre Specified Outcome: Implementation Climate Scale
Description: Implementation climate scale (Jacobs et al., 2014). This scale contains 6 items scored on a 1 to 5 scale. An average score across the 6 items will be calculated per provider. Possible scores on this outcome range from a minimum of 1 to a maximum of 6. Higher scores indicate a more positive implementation climate, which is a better outcome.
Time Frame: From baseline to 9 months post baseline
Population: Table reports means and standard deviations with listwise deletion. The pre-specified plan uses mixed models with full maximum likelihood estimation (intent-to-treat) and data from N=54 ATTC providers and N=58 E-ATTC providers.
Measure: Mean (Standard Deviation); unit: Units on Implementation Climate Scale
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Number analyzed (Participants) | 54 | 58
Units on Implementation Climate Scale | 3.77 (1.17) | 4.27 (0.81)
Statistical Analysis 1: Comparison: Addiction Technology Transfer Center (ATTC) Training vs Enhanced ATTC (E-ATTC) Training Strategy; These analyses are unadjusted. The primary outcomes paper will report both unadjusted and adjusted analyses; Test type: Superiority — Analyses are at the provider-level. Only those providers who completed the post-implementation survey (at the end of the 9-month implementation phase) were included in the analysis; p = .011, t-test, 2 sided — Means were compared between conditions in an independent-samples T-test; T-test adjusted for inequality of variances; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.88 to 0.12], Standard Error of Mean 0.191

7. Other Pre Specified Outcome: Leadership Engagement Scale
Description: Measure of leadership engagement (Garner, unpublished data). The scale contains 4 items scored on a 1 to 5 scale. An average perceived leadership engagement scale will be calculated for each provider. Possible scores on this outcome range from a minimum score of 1 to a maximum score of 5. Higher scores indicate higher perceived leadership engagement, which is a better outcome.
Time Frame: From baseline to 9 months post baseline
Population: Table reports means and standard deviations with listwise deletion. The pre-specified plan uses mixed models with full maximum likelihood estimation (intent-to-treat) and data from N=53 ATTC providers and N=58 E-ATTC providers.
Measure: Mean (Standard Deviation); unit: Units on Leadership Engagement Scale
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
Number analyzed (Participants) | 53 | 58
Units on Leadership Engagement Scale | 3.47 (1.27) | 3.75 (1.17)
Statistical Analysis 1: Comparison: Addiction Technology Transfer Center (ATTC) Training vs Enhanced ATTC (E-ATTC) Training Strategy; These analyses are unadjusted. The primary outcomes paper will report both unadjusted and adjusted analyses; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = .218, t-test, 2 sided — Means of leadership engagement scores were compared between conditions in an independent-samples T-test; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.75 to 0.17], Standard Error of Mean 0.232

ADVERSE EVENTS:
Time Frame: Adverse event data were collected as part of comprehensive follow-up assessments (twice over a 6-month period for patients and twice over a 9-month period for providers).
Description: Used standard National Institutes of Health definition of study-related adverse and serious adverse events.
  Adverse events and serious adverse events were assessed systematically as part of the comprehensive follow-up assessments.
Arm/Group | Addiction Technology Transfer Center (ATTC) Training | Enhanced ATTC (E-ATTC) Training Strategy
All-Cause Mortality (participants affected / at risk) | 1/381 | 1/399
Serious Adverse Events (participants affected / at risk) | 1/381 | 1/399
Other Adverse Events (participants affected / at risk) | 0/381 | 0/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Addiction Technology Transfer Center (ATTC) Training (N=381) | Enhanced ATTC (E-ATTC) Training Strategy (N=399)
Death (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Two participants lost to overdose over the follow up period (also recorded in the all-cause mortality section)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT03931174/Prot_SAP_001.pdf
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT03931174/ICF_002.pdf